CLINICAL TRIAL: NCT04447092
Title: Biomarker-oriented Study of Pembrolizumab in Combination With Chemotherapy in Chemotherapy -naïve Advanced Pancreatic Cancer
Brief Title: Pembrolizumab Plus Chemotherapy in 1st Line Treatment of Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2003-235-1115
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; pembrolizumab; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemcitabine/Nab-paclitaxel (Experimental): Gemcitabine/Nab-paclitaxel + pembrolizumab
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Pembrolizumab
- FOLFIRINOX (Experimental): FOLFIRINOX + pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5FU

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 iv D1, 8, 15 (every 4 weeks)
  Arms: Gemcitabine/Nab-paclitaxel
Drug: Nab-paclitaxel — Nab-paclitaxel 125 mg/m2 iv D1, 8, 15 (every 4 weeks)
  Arms: Gemcitabine/Nab-paclitaxel
Drug: Pembrolizumab — Pembrolizumab ( 200 ) mg iv D1 (every 3 weeks)
Drug: Oxaliplatin — Oxaliplatin 65 mg/m2 iv over 2 hours D1 (every 2 weeks)
  Arms: FOLFIRINOX
Drug: Leucovorin — Leucovorin 400 mg/m2 iv D1 (every 2 weeks)
  Arms: FOLFIRINOX
Drug: Irinotecan — Irinotecan 140 mg/m2 iv over 1.5 hours D1 (every 2 weeks)
  Arms: FOLFIRINOX
Drug: 5FU — 5-FU 2400 mg/m2 iv over 46 hours D1 (every 2 weeks)
  Arms: FOLFIRINOX

SUMMARY:
This is an open-label, phase 2 study of Pembrolizumab in combination with chemotherapy in chemotherapy-naïve advanced pancreatic cancer

DETAILED DESCRIPTION:
* In unresectable advanced pancreatic cancer, palliative chemotherapy (mainly Gemcitabine/nab-Paclitaxel or FOLFIRINOX) is the mainstay of treatment. Regardless of the choice of first-line therapy, more than half of the patients with advanced/metastatic disease will progress within six months and will not survive more than one year.
* Immune cells (IC) are a significant part of the pancreatic tumor-associated stroma and play a fundamental part in maintaining a non-immunogenic and immuno-suppressive environment.
* IO (Immuno-Oncology drug) monotherapy is not effective in advanced pancreatic cancer; therefore, we need more active combination regimens including IO/IO or IO/chemotherapy, etc. Furthermore, we need biomarker study to uncover which population is an optimal target for this IO-based treatment strategy.
* Based on these rationale, we plan to conduct an open-label, phase 2 study to explore biomarkers and evaluate the safety and efficacy of the pembrolizumab/chemotherapy combination in an advanced pancreatic cancer primary environment.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent
2. Histologically confirmed diagnosis of unresectable, recurrent, or metastatic pancreatic cancer
3. Not pregnant, not breasfeeding, and agree to use proper contraception,
4. Chemotherapy-naïve for advanced pancreatic cancer (previous adjuvant chemotherapy is allowed)
5. Have measurable disease based on RECIST 1.1.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Have adequate organ function

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) 1.5 (or 1.0) x (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>75,000 per mm3)
   * Serum creatinine CL>30 mL/min by the Cockcroft-Gault formula or serum creatinine ≤1.5 × ULN
   * Serum bilirubin ≤ 1.5 x ULN
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤ 5x ULN
   * International normalized ratio (INR) or Prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks
4. Has received prior radiotherapy within 2 weeks of start of study treatment.
5. Has received a live vaccine within 30 days prior to the first dose of study drug.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.
9. Has known active CNS metastases and/or carcinomatous meningitis.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV).
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 8 weeks
  The percentage of patients whose optimal response achieves CR or PR between the initial response assessment and the time between treatment termination or intermediate dropout due to any cause

SECONDARY OUTCOMES:
Progression-free survival | 8 weeks
  Time from enroll until disease progression or death
Duration of response | 8 weeks
  Time from enroll untill disease progression or death in patients whose optimal response achieves CR or PR
Disease control rate | 8 weeks
  The percentage of patients who have achieved complete response, partial response and stable disease
Overall survival | 8 weeks
  Time from enroll until death from any cause
Immune-related response | 8 weeks
  RECIST 1.1, ir response

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, M.D., PhD., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No